CLINICAL TRIAL: NCT05080127
Title: The Feasibility of Systemic Reaction After Contact Exposure to the Allergenic Food in Children With Known Food Allergy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, idit roth, Allergy and Immunology specialist, Meir Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0355-19-MMC
Record Dates: First submitted 2021-09-27; First posted 2021-10-15 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Food Allergy; Quality of Life
Keywords: food allergy; contact allergic reaction; skin prick test
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Intervention Model Description: * study group - 500 children with known food allergy
  * control groups - A. 50 children with atopic comorbidities but no food allergy. B. 50 children without atopic comorbidities
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- study subjects (Experimental): Children with proven IgE-mediated food allergy to one of the allergenic foods described.
  Parallel to the skin tests that are done as part of the accepted follow-up:
  1. The parents will fill a questionnaire regarding the quality of life (QOL) and another questionnaire regards family and personal relevant medical history.
  2. Patch test sticker with the allergenic food will be placed on the forearm for 15 minutes.
  3. A week later and 2 months later, the same QOL questionnaire will be sent by e-mail.
  Interventions: Combination Product: application of the allergenic food
- Control - atopic children (Active Comparator): Children with atopic comorbidities except for food allergy (ie. atopic dermatitis, asthma, allergic rhinitis).
  1. The parents will fill a questionnaire regarding family and personal relevant medical history and foods that the child is exposed to regularly.
  2. Patch test stickers with two of the food allergen list will be placed on the forearm for 15 minutes.
  Interventions: Combination Product: application of the allergenic food
- Control - healthy children (Active Comparator): Children without any atopic comorbidity (ie. atopic dermatitis, asthma, allergic rhinitis, and food allergy).
  1. The parents will fill a questionnaire regarding family and personal relevant medical history and foods that the child is exposed to regularly.
  2. Patch test stickers with two of the food allergen list will be placed on the forearm for 15 minutes.
  Interventions: Combination Product: application of the allergenic food

INTERVENTIONS:
Combination Product: application of the allergenic food — a small amount of the allergenic fresh food will be placed on the forearm using a patch test sticker for 15 minutes. the skin reaction will be measured.

SUMMARY:
The prevalence of food allergy in the western world is a growing health problem. The majority of reactions are caused due to oral exposure to the known food allergen. However, there are reports about allergic symptoms after exposure to the allergenic food by contact and/ or inhalation. Most of those reports are subjective without an objective report of healthcare professionals. There are only a few prospective studies that observed objectively the "reliability" of those subjective reports. The estimated chance for systemic allergic reaction due to skin prick test with fresh food is 0.008%, and even then it will not cause anaphylaxis that will need epinephrine use. That evidence is in concordance with our experience. Even with all the information gathered, a study that examines the chance of systemic reaction after skin contact with the allergenic food is still missing.

Additionally, lately, researchers start to examine the influence of food allergy on the quality of life (QOL) of allergic children and their parents. As expected, all studies show negative effects on QOL. The major concern of the parents is from random exposure and severe allergic reaction due to contact with the allergenic food. As far as the investigators know, no study examined the influence of supervised contact with allergenic food on the fear of the child and his parents.

The study aims to evaluate the risk for a systemic allergic reaction after skin exposure to allergenic food in children with known food allergy.

DETAILED DESCRIPTION:
The prevalence of food allergy in the western world is estimated at 8% and is constantly raising. The majority of reactions are caused due to oral exposure to the known food allergen. However, there are reports about allergic symptoms after exposure to the allergenic food by contact and/ or inhalation. Most of those reports are subjective without an objective report of a healthcare professional. There is one description of a 16-year-old boy with cow's milk allergy (CMA), who developed anaphylaxis from skin exposure to small amount of cow's milk under the supervision of a healthcare professional. There are only a few prospective studies that observed objectively the "reliability" of those subjective reports. In 2003, Simonte SJ et al examine 30 children with known peanut allergy of which 19 reported past reactions after contact/ inhaled exposure to peanuts. They did a supervised exposure to contact and inhalation of peanut butter. They reported only local skin reactions such as redness (10%), itching (17%), and wheal and flare (7%) with no systemic reactions. Other studies examine the allergic reactions to skin contact with peanuts and also did not report on systemic reactions. In one of the studies they examine the allergic reaction to skin contact in 330 children allergic to peanuts and only 41% had a local reaction with no systemic reactions. In the second study, the investigators did the accepted skin prick test (SPT) with peanut and immediate skin application food test (I-SAFT) with peanut butter in 84 children. The investigators did not observe systemic allergic reactions. Only one study examined allergic reactions after contact with cow's milk in children with CMA. The aim of this study was to compare the skin reaction of children with CMA with and without atopic dermatitis (AD). The investigators did not report systemic reactions also. There are few cases reports that described systemic allergic reaction during SPT, all cases were with fish allergy. A large study examined reactions to SPT with fresh food on 1,138 allergic patients. The investigators have shown that the chance of systemic allergic reaction is 0.008%, and none of the cases needed epinephrine. They review other 15 studies and did not find evidence to systemic reaction after SPT except for one study that reported a 0.005% prevalence of systemic reaction to follow SPT with fresh food in infants younger than 6 months of age.

That evidence is in concordance with the investigators experience. Until today, the investigators did not see the systemic reaction after SPT in children with food allergies. Even with all the information gathered, a study that examines the chance of systemic reaction after skin contact with the allergenic food is still missing.

Additionally, lately, researchers start to examine the influence of food allergy on the quality of life (QOL) of allergic children and their parents. As expected, all studies show a negative effect on QOL. The major concern of the parents is from random exposure and severe allergic reaction due to contact with the allergenic food. As far as the investigator know, no study examined the influence of supervised contact with allergenic food on the fear of the child and his parents.

The study aims primarily - to evaluate the risk for a systemic allergic reaction after skin exposure to the allergenic food in children with known food allergies.

secondary - 1. To evaluate the QOL of the parents (and children over 8 years) before and after the contact with the allergenic food.

Methods: 500 children with known food allergy and 100 children without food allergy as a control group. Simultaneously to the regular skin prick tests, a patch test sticker with the allergenic food will be placed on the forearm for 15 minutes. The parents will fill quality of life questionnaire before the tests, a week later, and 2 months later.

expected results - No allergic reaction will occur after the patch test other than mild local reaction. the level of anxiety will be reduced after the tests.

ELIGIBILITY:
Inclusion Criteria:

* Children aged one year to 18 years old with proven food allergy to one of the foods mentioned above.

Exclusion Criteria:

* under 12 months of age
* Admitted in the past in intensive care unit after allergic reaction
* Had allergic reaction that treated with three or more adrenalin doses (EpiPen/ IM adrenaline)
* Uncontrolled asthma (according to the GINA guidelines)
* Severe AD
* Children with allergy to three or more allergens not from the same allergen group

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
reaction to the patch test | 15 minutes
  systemic or local reaction after the skin test with the patch test

SECONDARY OUTCOMES:
change in quality of life | 2 months
  change in the perception of qality of life by the parents after a week and two months from the tests compared to qality of life questionnaire before the test.
  Quality of life scale is 0-84 and the highest the score the quality of life is lower.

CONTACTS AND LOCATIONS:
Overall Officials: Idit Lachover- Roth, MD, Principal Investigator — Meir Medical Center
Locations (2):
- Israel (2):
  - Allergy and Clinical Immunology Unit, Kfar Saba
  - Meir medical center, Kfar Saba

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sicherer SH, Sampson HA. Food allergy: Epidemiology, pathogenesis, diagnosis, and treatment. J Allergy Clin Immunol. 2014 Feb;133(2):291-307; quiz 308. doi: 10.1016/j.jaci.2013.11.020. Epub 2013 Dec 31. PMID 24388012
- [Background] Dominguez C, Ojeda I, Crespo JF, Pascual C, Ojeda A, Martin-Esteban M. Allergic reactions following skin contact with fish. Allergy Asthma Proc. 1996 Mar-Apr;17(2):83-7. doi: 10.2500/108854196778645092. PMID 8934799
- [Background] McIntyre CL, Sheetz AH, Carroll CR, Young MC. Administration of epinephrine for life-threatening allergic reactions in school settings. Pediatrics. 2005 Nov;116(5):1134-40. doi: 10.1542/peds.2004-1475. PMID 16264000
- [Background] Sicherer SH, Furlong TJ, DeSimone J, Sampson HA. The US Peanut and Tree Nut Allergy Registry: characteristics of reactions in schools and day care. J Pediatr. 2001 Apr;138(4):560-5. doi: 10.1067/mpd.2001.111821. PMID 11295721
- [Background] Liccardi G, De Falco F, Gilder JA, D'Amato M, D'Amato G. Severe systemic allergic reaction induced by accidental skin contact with cow milk in a 16-year-old boy. A case report. J Investig Allergol Clin Immunol. 2004;14(2):168-71. PMID 15301310
- [Background] Dinakar C, Shroba J, Portnoy JM. The transforming power of proximity food challenges. Ann Allergy Asthma Immunol. 2016 Aug;117(2):135-7. doi: 10.1016/j.anai.2016.06.015. No abstract available. PMID 27499540
- [Background] Schichter-Konfino V, Almog M, Bamberger E, Berkowitz D, Kessel A. The significance of allergic contact urticaria to milk in children with cow's milk allergy. Pediatr Allergy Immunol. 2015 May;26(3):218-222. doi: 10.1111/pai.12375. PMID 25775957
- [Background] Simonte SJ, Ma S, Mofidi S, Sicherer SH. Relevance of casual contact with peanut butter in children with peanut allergy. J Allergy Clin Immunol. 2003 Jul;112(1):180-2. doi: 10.1067/mai.2003.1486. PMID 12847496
- [Background] Wainstein BK, Kashef S, Ziegler M, Jelley D, Ziegler JB. Frequency and significance of immediate contact reactions to peanut in peanut-sensitive children. Clin Exp Allergy. 2007 Jun;37(6):839-45. doi: 10.1111/j.1365-2222.2007.02726.x. PMID 17517097
- [Background] Wainstein BK, Yee A, Jelley D, Ziegler M, Ziegler JB. Combining skin prick, immediate skin application and specific-IgE testing in the diagnosis of peanut allergy in children. Pediatr Allergy Immunol. 2007 May;18(3):231-9. doi: 10.1111/j.1399-3038.2007.00517.x. PMID 17433001
- [Background] Pitsios C, Dimitriou A, Kontou-Fili K. Allergic reactions during allergy skin testing with food allergens. Eur Ann Allergy Clin Immunol. 2009 Aug;41(4):126-8. PMID 19877567
- [Background] Pitsios C, Dimitriou A, Stefanaki EC, Kontou-Fili K. Anaphylaxis during skin testing with food allergens in children. Eur J Pediatr. 2010 May;169(5):613-5. doi: 10.1007/s00431-009-1070-5. Epub 2009 Sep 23. PMID 19771451
- [Background] Codreanu F, Moneret-Vautrin DA, Morisset M, Guenard L, Rance F, Kanny G, Lemerdy P. The risk of systemic reactions to skin prick-tests using food allergens: CICBAA data and literature review. Eur Ann Allergy Clin Immunol. 2006 Feb;38(2):52-4. PMID 16711536
- [Background] Devenney I, Falth-Magnusson K. Skin prick tests may give generalized allergic reactions in infants. Ann Allergy Asthma Immunol. 2000 Dec;85(6 Pt 1):457-60. doi: 10.1016/S1081-1206(10)62571-9. PMID 11152165
- [Background] DunnGalvin A, Dubois AE, Flokstra-de Blok BM, Hourihane JO. The effects of food allergy on quality of life. Chem Immunol Allergy. 2015;101:235-52. doi: 10.1159/000375106. Epub 2015 May 21. PMID 26022884